CLINICAL TRIAL: NCT01040416
Title: Endoscopic Therapy for Actively Bleeding Marginal Ulcers: Our Experience After 7,020 Roux-en-Y Gastric Bypass Surgeries
Brief Title: Endoscopic Therapy for Bleeding Marginal Ulcers After Gastric Bypass
Acronym: BleedingMU
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Kelvin D Higa, MD; FACS; FASMBS; Professor of Surgery, University of California San Francisco, UCSF Fresno / ALSA Medical Group, Inc. Minimally Invasive Surgery Program
Other Study IDs: CMC IRB No. 2008081; U1111-1112-9849 (Other: World Health Organization, Universal Trial Number)
Record Dates: First submitted 2009-12-23; First posted 2009-12-29 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-12

CONDITIONS: Bleeding Marginal Ulcer
Keywords: complicated marginal ulcer; complex marginal ulcer; complication after gastric bypass; gastrointestinal hemorrhage
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Bleeding marginal ulcer after RYGB

SUMMARY:
The objective of this study is to identify the incidence rate; describe the risk factors, clinical presentation, and endoscopic treatment; assess the morbidity, mortality, and overall performance of the management of patients with actively bleeding marginal ulcers after Roux-en-Y gastric bypass (RYGB) surgery.

DETAILED DESCRIPTION:
Marginal ulceration "MU", which presents as an ulcer at the margins of the gastrojejunostomy on the jejunal side, is a common late complication after RYGB. Its incidence after RYGB ranges from as low as 0.6 to as high as 16%. In our hands with the laparoscopic hand-sewn technique for the GJ, the incidence is 1.4%. The presence of specific technical factors - staple-line dehiscence or gastro-gastric fistula, enlarged pouch, foreign material and local ischemia - and environmental factors - tobacco, NSAID´s, alcohol consumption, and H pylori infection among others - have been associated with marginal ulceration however the exact etiopathogenesis has not been completely elucidated.

Similar to peptic ulcer disease (PUD), most marginal ulcers respond to medical therapy, specifically sucralfate and acid-lowering medication. In contrast, complicated marginal ulcers - perforation, bleeding, or chronicity (obstruction, penetration, and intractability)- warrants operative intervention.

Early presentation of hemorrhage after RYGB is mostly related to staple-line failure and may result in either GI or intraabdominal hemorrhage. When indicated, operative interventions consist of either endoscopic therapy, re-operation, or both. In contrast, late presentation of gastrointestinal hemorrhage after RYGB is mostly secondary to a bleeding marginal ulcer however complicated peptic ulcer disease can present in the excluded stomach and duodenum as well.

Most literature available for the management of GI hemorrhage after RYGB is for the early presentation of hemorrhage secondary to staple-line failure. Hence, options for endoscopic hemostatic therapy described in this scenario are I) injection therapy, II) coagulation therapy, III) endoscopic clipping, and IV) a combined modality (for example injection & coagulation or injection and clipping).

The feasibility, reliability, reproducibility, efficacy, validity and safety of the endoscopic hemostatic therapy for acutely bleeding peptic ulcers has been well documented. Multiple risk-stratification tools for upper-GI hemorrhage have also been developed such as the Blatchford, clinical and complete Rockall scores, and the Forrest classification. Moreover, pre and post endoscopic schemes of PPI´s therapy in patients with bleeding peptic ulcers is effective and cost-saving. However, All of them have not been validated in the obese population status post RYGB complicated with a bleeding marginal ulcer.

Summarizing, there is scant information about the management of late complications after gastric bypass especially after the widespread adoption of the laparoscopic approach and the modern anatomical construct of Roux-en-Y Gastric Bypass surgery. We formally analyze the management efficacy of patients with actively bleeding marginal ulcers after Roux-en-Y gastric bypass (RYGB) surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients status post laparoscopic RYGB surgery with active gastrointestinal hemorrhage secondary to marginal ulcer

Exclusion Criteria:

* bleeding marginal ulcers after other bariatric procedures
* staple-line bleeding after RYGB
* iron-deficiency anemia (chronic) secondary to non-actively bleeding marginal ulcer after RYGB
* other sources of GI bleeding different from marginal ulcer such as from staple-lines, complicated PUD, and other surgical and medical causes of GI hemorrhage
* missing records and/or unreachable patients with scant information for analysis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with actively bleeding marginal ulcers after Roux-en-Y gastric bypass (RYGB) surgery.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Morbidity and mortality, overall | throughout follow-up
re-bleeding, gastrointestinal hemorrhage secondary to marginal ulceration | throughout follow-up
marginal ulcer recurrence | at last follow-up
Symptom resolution, marginal ulcer | at last follow-up

SECONDARY OUTCOMES:
consumption of blood products | during bleeding-related hospitalization
weight loss expressed as Body Mass Index and Percentage excess weight loss | at the lowest point and yearly intervals

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Tercero, MD, Study Director — Research Associate, University of California San Francisco; Kelvin D Higa, MD, Principal Investigator — Professor of Surgery, University of California San Francisco
Locations (1):
- UCSF Fresno Center for Medical Education and Research, Fresno, California, United States

REFERENCES:
- [Background] Higa KD, Boone KB, Ho T, Davies OG. Laparoscopic Roux-en-Y gastric bypass for morbid obesity: technique and preliminary results of our first 400 patients. Arch Surg. 2000 Sep;135(9):1029-33; discussion 1033-4. doi: 10.1001/archsurg.135.9.1029. PMID 10982506
- [Background] Hedley AA, Ogden CL, Johnson CL, Carroll MD, Curtin LR, Flegal KM. Prevalence of overweight and obesity among US children, adolescents, and adults, 1999-2002. JAMA. 2004 Jun 16;291(23):2847-50. doi: 10.1001/jama.291.23.2847. PMID 15199035
- [Background] McTigue KM, Harris R, Hemphill B, Lux L, Sutton S, Bunton AJ, Lohr KN. Screening and interventions for obesity in adults: summary of the evidence for the U.S. Preventive Services Task Force. Ann Intern Med. 2003 Dec 2;139(11):933-49. doi: 10.7326/0003-4819-139-11-200312020-00013. PMID 14644897
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Christou NV, Sampalis JS, Liberman M, Look D, Auger S, McLean AP, MacLean LD. Surgery decreases long-term mortality, morbidity, and health care use in morbidly obese patients. Ann Surg. 2004 Sep;240(3):416-23; discussion 423-4. doi: 10.1097/01.sla.0000137343.63376.19. PMID 15319713
- [Background] Adams TD, Gress RE, Smith SC, Halverson RC, Simper SC, Rosamond WD, Lamonte MJ, Stroup AM, Hunt SC. Long-term mortality after gastric bypass surgery. N Engl J Med. 2007 Aug 23;357(8):753-61. doi: 10.1056/NEJMoa066603. PMID 17715409
- [Background] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Background] Cremieux PY, Buchwald H, Shikora SA, Ghosh A, Yang HE, Buessing M. A study on the economic impact of bariatric surgery. Am J Manag Care. 2008 Sep;14(9):589-96. PMID 18778174
- [Background] Santry HP, Gillen DL, Lauderdale DS. Trends in bariatric surgical procedures. JAMA. 2005 Oct 19;294(15):1909-17. doi: 10.1001/jama.294.15.1909. PMID 16234497
- [Background] Flum DR, Khan TV, Dellinger EP. Toward the rational and equitable use of bariatric surgery. JAMA. 2007 Sep 26;298(12):1442-4. doi: 10.1001/jama.298.12.1442. No abstract available. PMID 17895461
- [Background] Meguid MM, Glade MJ, Middleton FA. Weight regain after Roux-en-Y: a significant 20% complication related to PYY. Nutrition. 2008 Sep;24(9):832-42. doi: 10.1016/j.nut.2008.06.027. PMID 18725080
- [Background] Nguyen NT. Reoperations and revisions in bariatric surgery. Surg Endosc. 2007 Nov;21(11):1907-8. doi: 10.1007/s00464-007-9572-6. Epub 2007 Sep 8. No abstract available. PMID 17828427
- [Background] Sapala JA, Wood MH, Sapala MA, Flake TM Jr. Marginal ulcer after gastric bypass: a prospective 3-year study of 173 patients. Obes Surg. 1998 Oct;8(5):505-16. doi: 10.1381/096089298765554061. PMID 9819081
- [Background] Higa KD, Boone KB, Ho T. Complications of the laparoscopic Roux-en-Y gastric bypass: 1,040 patients--what have we learned? Obes Surg. 2000 Dec;10(6):509-13. doi: 10.1381/096089200321593706. PMID 11175957
- [Background] Sanyal AJ, Sugerman HJ, Kellum JM, Engle KM, Wolfe L. Stomal complications of gastric bypass: incidence and outcome of therapy. Am J Gastroenterol. 1992 Sep;87(9):1165-9. PMID 1519574
- [Background] Capella JF, Capella RF. Staple Disruption and Marginal Ulceration in Gastric Bypass Procedures for Weight Reduction. Obes Surg. 1996 Feb;6(1):44-49. doi: 10.1381/096089296765557259. PMID 10731249
- [Background] Capella JF, Capella RF. Gastro-gastric fistulas and marginal ulcers in gastric bypass procedures for weight reduction. Obes Surg. 1999 Feb;9(1):22-7; discussion 28. doi: 10.1381/096089299765553674. PMID 10065576
- [Background] Jordan JH, Hocking MP, Rout WR, Woodward ER. Marginal ulcer following gastric bypass for morbid obesity. Am Surg. 1991 May;57(5):286-8. PMID 2039124
- [Background] Sacks BC, Mattar SG, Qureshi FG, Eid GM, Collins JL, Barinas-Mitchell EJ, Schauer PR, Ramanathan RC. Incidence of marginal ulcers and the use of absorbable anastomotic sutures in laparoscopic Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2006 Jan-Feb;2(1):11-6. doi: 10.1016/j.soard.2005.10.013. PMID 16925306
- [Background] Lublin M, McCoy M, Waldrep DJ. Perforating marginal ulcers after laparoscopic gastric bypass. Surg Endosc. 2006 Jan;20(1):51-4. doi: 10.1007/s00464-005-0325-0. Epub 2005 Dec 7. PMID 16333541
- [Background] St Jean MR, Dunkle-Blatter SE, Petrick AT. Laparoscopic management of perforated marginal ulcer after laparoscopic Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2006 Nov-Dec;2(6):668. doi: 10.1016/j.soard.2006.09.011. No abstract available. PMID 17138240
- [Background] Chin EH, Hazzan D, Sarpel U, Herron DM. Multimedia article. Laparoscopic repair of a perforated marginal ulcer 2 years after gastric bypass. Surg Endosc. 2007 Nov;21(11):2110. doi: 10.1007/s00464-007-9486-3. Epub 2007 Aug 18. PMID 17704879
- [Background] Wheeler AA, de la Torre RA, Fearing NM. Laparoscopic repair of perforated marginal ulcer following Roux-en-Y gastric bypass: a case series. J Laparoendosc Adv Surg Tech A. 2011 Jan-Feb;21(1):57-60. doi: 10.1089/lap.2010.0402. Epub 2011 Jan 19. PMID 21247305
- [Background] Nguyen NT, Hinojosa MW, Gray J, Fayad C. Reoperation for marginal ulceration. Surg Endosc. 2007 Nov;21(11):1919-21. doi: 10.1007/s00464-007-9538-8. Epub 2007 Aug 19. No abstract available. PMID 17705072
- [Background] Patel RA, Brolin RE, Gandhi A. Revisional operations for marginal ulcer after Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2009 May-Jun;5(3):317-22. doi: 10.1016/j.soard.2008.10.011. Epub 2008 Nov 6. PMID 19136312
- [Background] Harnisch MC, Portenier DD, Pryor AD, Prince-Petersen R, Grant JP, DeMaria EJ. Preoperative weight gain does not predict failure of weight loss or co-morbidity resolution of laparoscopic Roux-en-Y gastric bypass for morbid obesity. Surg Obes Relat Dis. 2008 May-Jun;4(3):445-50. doi: 10.1016/j.soard.2007.09.016. PMID 18501309
- [Background] Madan AK, DeArmond G, Ternovits CA, Beech DJ, Tichansky DS. Laparoscopic revision of the gastrojejunostomy for recurrent bleeding ulcers after past open revision gastric bypass. Obes Surg. 2006 Dec;16(12):1662-8. doi: 10.1381/096089206779319400. PMID 17217644
- [Background] Nguyen NT, Longoria M, Chalifoux S, Wilson SE. Gastrointestinal hemorrhage after laparoscopic gastric bypass. Obes Surg. 2004 Nov-Dec;14(10):1308-12. doi: 10.1381/0960892042583879. PMID 15603643
- [Background] Nguyen NT, Hinojosa MW, Gray J et al. (2008). Gastrointestinal bleeding after Roux-en-Y gastric bypass. In Weight loss surgery: A multidisciplinary approach (pp. 401-4). Edgemont, PA: Matrix Medical Communications.
- [Background] Braley SC, Nguyen NT, Wolfe BM. Late gastrointestinal hemorrhage after gastric bypass. Obes Surg. 2002 Jun;12(3):404-7. doi: 10.1381/096089202321088255. PMID 12082897
- [Background] Gutthann SP, Garcia Rodriguez LA, Raiford DS. Individual nonsteroidal antiinflammatory drugs and other risk factors for upper gastrointestinal bleeding and perforation. Epidemiology. 1997 Jan;8(1):18-24. doi: 10.1097/00001648-199701000-00003. PMID 9116088
- [Background] Gralnek IM, Barkun AN, Bardou M. Management of acute bleeding from a peptic ulcer. N Engl J Med. 2008 Aug 28;359(9):928-37. doi: 10.1056/NEJMra0706113. No abstract available. PMID 18753649
- [Background] Barkun AN. Should every patient with suspected upper GI bleeding receive a proton pump inhibitor while awaiting endoscopy? Gastrointest Endosc. 2008 Jun;67(7):1064-6. doi: 10.1016/j.gie.2008.02.040. No abstract available. PMID 18513549
- [Background] Fernandez-Esparrach G, Bordas JM, Pellise M, Gimeno-Garcia AZ, Lacy A, Delgado S, Cardenas A, Gines A, Sendino O, Momblan D, Zabalza M, Llach J. Endoscopic management of early GI hemorrhage after laparoscopic gastric bypass. Gastrointest Endosc. 2008 Mar;67(3):552-5. doi: 10.1016/j.gie.2007.10.024. PMID 18294521
- See also: "Click here for more information about the department sponsor´s web site" — http://www.fresno.ucsf.edu/surgery